CLINICAL TRIAL: NCT04771039
Title: Ocular Manifestations of Chronic Inflammatory Bowel Disease (IBD): Retrospective Study in the Hepato-gastroenterology Department of the Nancy CHRU
Brief Title: Ocular Manifestations of Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: HRIPH
Record Dates: First submitted 2021-01-04; First posted 2021-02-25 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2020-12

CONDITIONS: Inflammatory Bowel Diseases; Ophthalmopathy
MeSH Terms: conditions — Inflammatory Bowel Diseases; Eye Diseases | interventions — Referral and Consultation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with chronic inflammatory bowel disease who consulted in ophthalmology
  Interventions: Other: reason for consultation

INTERVENTIONS:
Other: reason for consultation — search in medical files for reasons for ophthalmology consultation, functional signs, clinical signs, treatment, characteristics of IBD

SUMMARY:
Ocular damage is found in the 3rd rank of extra intestinal manifestations (MEI) Potentially serious functional complications (see uveitis and risk of blindness) requiring rapid management Rare uveitis in the literature (0.5% -3%), study on a large sample to assess their prevalence in patients with IBD at the Nancy CHRU and describe all the ocular manifestations that can be found.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients followed at Nancy University Hospital for IBD and having consulted in the ophthalmology department

Exclusion Criteria:

* Minor patients
* patients without IBD
* patients for whom there is no ophthalmology consultation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients followed at Nancy University Hospital for IBD and having consulted in the ophthalmology department
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-12 (Actual)

PRIMARY OUTCOMES:
frequency | baseline
  frequency of ocular manifestations in inflammatory bowel disease

SECONDARY OUTCOMES:
Number | baseline
  Number of uveitis, scleritis and episcleritis; prevalence calculation

IPD SHARING:
Plan to Share IPD: Undecided